CLINICAL TRIAL: NCT02963012
Title: The Correlation Between Uterine Endometrial Pattern and Ectopic Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Ziv Medical Center (Other)
Responsible Party: Principal Investigator, Etty Spiegel, head of ultrasound unit, HaEmek Medical Center, Israel
Other Study IDs: emc 0164-15
Record Dates: First submitted 2016-09-12; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ultrasound examination

SUMMARY:
A prospective trail. Pregnant women in the first trimester with positive BHCG and no visualization of gestational sac will be recruited.

The correlation between endometrial pattern and ectopic pregnancy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* First trimester of pregnancy
* No visualization of gestational sac

Exclusion Criteria:

* Hemodynamic instability

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with ectopic pregnancy, in the first trimester.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the corellation between presence and width of trilaminar endometrium as evaluated by transvaginal ultrasound and the diagnosis of ectopic pregnancy | first trimester of pregnancy

IPD SHARING:
Plan to Share IPD: Undecided